CLINICAL TRIAL: NCT01096836
Title: Combined Effects of Resistance Training and Low Carbohydrate or Conventional Diets on Strength, Muscle Mass, Body Composition, Blood Lipids and Endothelium Function
Brief Title: Low Carbohydrate and Conventional Diets Associated to Resistance Training on Muscle Fitness and Health Markers
Acronym: LCD-RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Gama Filho (Other)
Responsible Party: Prof. Paulo Sergio Chagas Gomes, Ph.D., Universidade Gama Filho
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UGF-01-2010
Record Dates: First submitted 2010-03-17; First posted 2010-03-31 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2007-11

CONDITIONS: Obesity; Overweight
Keywords: resistance exercise; body mass index; hypertrophy; endothelial function; blood lipids
MeSH Terms: conditions — Obesity; Overweight; Hypertrophy | interventions — Nutrients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet counseling (Experimental): Outcomes of the study may enhance diet counseling
  Interventions: Other: macronutrient and energy manipulation
- exercise training (Experimental)
  Interventions: Other: macronutrient and energy manipulation

INTERVENTIONS:
Other: macronutrient and energy manipulation

SUMMARY:
The purpose of this study was to compare the effects of two different diets (low carbohydrate - LCD and conventional - CONV) on body composition, strength performance, muscle mass and biomarkers of health in overweight adults submitted to resistance training (RT). It has been hypothesized that LCD would produce higher rates of weight loss and that both diets would be useful to maintain muscle mass and strength and biomarkers of health.

DETAILED DESCRIPTION:
Overweight and obesity prevalence has increased worldwide. Current guidelines recommend health behavior modifications, including better eating habits and regular physical activity (including resistance training - RT) as a strategy to control and prevent the problem. Traditionally, diets poor in energy and fat (conventional diets - CONV) have been recommended to promote losses in body and fat masses; however, there has been recently a growing interest in the academic community to investigate the effects of low carbohydrate diet (LCD) on health outcomes, since this kind of diet appears to be more effective for reducing body mass as compared to CONV. Nevertheless, evidences are scarce regarding the effects of LCD associated to RT on body composition, strength performance, blood lipids, endothelium function and other markers of health, demanding the development of clinical trials aiming to determine the combined health effects of these interventions.

ELIGIBILITY:
Inclusion Criteria:

* BMI equal or over 25 kg/m2
* resistance trained at least 12 weeks

Exclusion Criteria:

* upper or lower limbs injury
* pregnancy
* diabetes
* use of ergogenics, stimulants or drugs
* history of dislipidemias
* arterial hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2006-09; Primary Completion 2008-01 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
body mass | eight weeks
  Measured always at the same time of the day on a calibrated weight scale

SECONDARY OUTCOMES:
Muscle strength | eight weeks
  Measured using resistance exercise machines (isotonic) in four exercise movements
Endothelial function | eight weeks
  Measured using a two dimensional color spectral Doppler ultrasound equipped with a 14MHz linear transducer. Subject laid down comfortably in the supine position with the right arm slightly abduced. After locating the brachial artery, the transducer was placed on the anteromedial face of the right arm, perpendicular to the centerline of the arm, 5-10 cm above the antecubital fossa, over the artery.
muscle thicknesses | eight weeks
  Measured with a ultrasoundo bidimensional in Mode B, with a 7,5MHz transducer on the anatomical sites knee extensor muscles and elbow flexors and extensors.
markers of renal function | eight weeks
  Measured using conventional and satandardized laboratory methods with subjects fasting for 12 hours
body composition | eight weeks
  Measured with skinfold calipers and using prediction equations to determine body fat and lean body mass.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Sergio C Gomes, Ph.D., Principal Investigator — Universidade Gama Filho
Locations (1):
- Laboratory Crossbridges, Rio de Janeiro, Rio de Janeiro, Brazil